CLINICAL TRIAL: NCT02603731
Title: Delirium at the Intensive Care Unit - a Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Stine Estrup, Junior Doctor, Zealand University Hospital
Other Study IDs: SE-DELIR1-15
Record Dates: First submitted 2015-11-04; First posted 2015-11-13 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Delirium; Intensive Care Unit Syndrome
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project seeks to describe the incidence of delirium in the Intensive Care Unit (ICU) and to identify risk and preventive factors associated with development of delirium.

Especially, the investigators want to investigate if an imitated natural light/dark cycle influences frequency of delirium.

DETAILED DESCRIPTION:
A common problem for patients in the ICU is episodes of delirium. Recent trials have described incidences ranging from 60-87% of patients in a number of different countries. Delirium is a condition with fluctuating conscience, disorganized thinking and disturbance of the sleep/wake cycle. Many patients with delirium experience hallucinations and agitation which can be very unpleasant for both patients and their families.

Some risk factors for the development of delirium well known, e.g. dementia, hypertension, illness severity (SAPS II score), delirium on the previous day, mechanical ventilation, emergency surgery and metabolic acidosis. The effect of sedative drug administration is not clear, as studies has been inconclusive.

Even though studies regarding the impact of sleep deprivation on development of delirium have been inconclusive, there is no doubt that delirious patients have a disturbed sleep-wake cycle, sleep architecture and circadian rhythm.

At the intensive care unit at the Department of Anesthesiology at Køge Hospital, three out of nine rooms have a simulated circadian light installed. The idea is that this light rhythm may help to keep a natural circadian rhythm, minimizing the risk of delirium.

With this descriptive and retrospective cohort study, the investigators therefore want to describe the incidence and possible risk- and preventive factors of delirium for the participants (ICU patients at Køge Hospital), and with a special focus on the possible effect of imitated circadian light..

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age admitted to the ICU at Køge Hospital in the study period

Exclusion Criteria:

* Richmond Agitation Sedation Score (RASS): -4 or -5 during the whole study period
* No CAM-ICU scores during the ICU stay
* Unable to communicate in Danish (aphasic, deaf, non-Danish speaking, severe brain damage)
* Severe dementia documented in electronic patient charts (OPUS)
* Patients not receiving active treatment (moribund patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU at Køge Hospital in the study period
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Delirium at any time point | Throughout study period, up to 6 months
  Incidence of patients with delirium during ICU-stay defined as at least one positive Confusion Assessment Method for the ICU (CAM-ICU) score or CAM-ICU negative delirium treated with anti-psychotics.

SECONDARY OUTCOMES:
Days with delirium | Throughout study period, up to 6 months
  Days with positive CAM-ICU or CAM-ICU negative delirium treated with anti-psychotics in relation to length of stay (LOS)
Circadian light exposure | Throughout study period, up to 6 months
  Difference in incidences of delirium between patients admitted to rooms with circadian rhythm lighting and standard rooms
Delirium in patients treated with hypnotics | Throughout study period, up to 6 months
  Difference in incidence of delirium in patients treated with hypnotics before admission to hospital (ATC N05C) compared to those who are not
Delirium in patients treated with steroids | Throughout study period, up to 6 months
  Differences in incidences of delirium in patients that are treated with systemic steroids vs. no treatment
Mortality | Throughout study period, up to 6 months
  Mortality within ICU stay
Demographic differences | Throughout study period, up to 6 months
  Incidence of delirium associated to demographic variables (age, gender)
Delirium and Simplified Acute Physiology Score (SAPS) | Throughout study period, up to 6 months
  Incidence of delirium associated to Simplified Acute Physiology Score (SAPS) II
Delirium related to number of ventilator days | Throughout study period, up to 6 months
  Incidence of delirium associated to number of ventilator days
Delirium related to sedation | Throughout study period, up to 6 months
  Incidence of delirium associated to sedation infusion
Delirium related to admission type | Throughout study period, up to 6 months
  Incidence of delirium associated to admission type (medical/elective surgical/acute surgical)
Distribution of types of delirium | Throughout study period, up to 6 months
  Incidence and distribution of delirium subtypes (hypoactive/hyperactive/mixed)

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mathiesen, MD, PhD, Study Chair — Køge Hospital
Locations (1):
- Køge Sygehus, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Svenningsen H, Tonnesen EK, Videbech P, Frydenberg M, Christensen D, Egerod I. Intensive care delirium - effect on memories and health-related quality of life - a follow-up study. J Clin Nurs. 2014 Mar;23(5-6):634-44. doi: 10.1111/jocn.12250. Epub 2013 May 6. PMID 23647511
- [Background] Girard TD, Jackson JC, Pandharipande PP, Pun BT, Thompson JL, Shintani AK, Gordon SM, Canonico AE, Dittus RS, Bernard GR, Ely EW. Delirium as a predictor of long-term cognitive impairment in survivors of critical illness. Crit Care Med. 2010 Jul;38(7):1513-20. doi: 10.1097/CCM.0b013e3181e47be1. PMID 20473145